CLINICAL TRIAL: NCT00866190
Title: A Phase 1B, Randomized, Placebo-Controlled, Double-Blinded, Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of Single-Daily Doses of SQ109 in Normal, Healthy Male and Female Volunteers
Brief Title: Dose Escalation Study of SQ109 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-0048; N01AI80024C; SQ-109
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-10

CONDITIONS: TB Multi-drug Resistant
Keywords: Mycobacterium tuberculosis, SQ109

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cohort 1 (Experimental): SQ109 dose 75 mg or placebo once daily for 14 days.
  Interventions: Drug: SQ109; Drug: Placebo
- Cohort 3 (Experimental): SQ109 dose 150 mg or placebo once daily for 14 days.
  Interventions: Drug: SQ109; Drug: Placebo
- Cohort 2 (Experimental): SQ109 dose 150 mg or placebo once daily on Days 1-5, 9, and 14.
  Interventions: Drug: SQ109; Drug: Placebo

INTERVENTIONS:
Drug: SQ109 — SQ109 150 mg is an oval, coated, white, scored tablet. Dosages: 75 mg administered once daily for 14 days; 150 mg administered once daily on Days 1-5, 9, and 14; and 150 mg administered once daily for 14 days.
Drug: Placebo — Placebo is an oval, coated, white, scored tablet administered once daily for 14 days or on Days 1-5, 9, and 14.

SUMMARY:
The purposes of this study are to determine: how safe it is to take SQ109 (an experimental tuberculosis treatment) once a day by mouth for up to 2 weeks in 2 different dosages; how well the body accepts it; how SQ109 enters and leaves the body and blood tissues over time; the amounts that can be detected in the blood; and how long it stays in the body. The study involves 30 volunteers: 24 will receive SQ109 and 6 will receive placebo (inactive substance). Qualified participants will be admitted to the study unit within 28 days from the screening and stay as inpatient for approximately 2 weeks. During this period they will receive study drug and complete all scheduled procedures including multiple blood draws. After discharge, there is a 14 day follow up period. Total study participation is about 56 days.

DETAILED DESCRIPTION:
Tuberculosis (TB) is one of the most important global health problems. According to recent estimates from the World Health Organization, 8 million new cases of TB and 1.9 million deaths from TB occur annually, making TB the second leading cause of death from an infectious pathogen. Due to multidrug resistant TB, the need for new and more effective drugs to treat TB is well recognized. This study is a phase 1B, prospective, single-center, double-blinded, randomized, placebo-controlled, clinical study of SQ109 to evaluate single-daily dose tolerability and pharmacokinetics (PK) of oral SQ109 in healthy subjects. The objectives of the study are to: determine the safety and tolerability of SQ109 administered daily for 14 days in healthy male and female volunteers; assess single dose and multiple dose PK of SQ109 administered daily for 14 days in healthy male and female volunteers; and assess single dose and multiple dose PK of SQ109 administered twice per week after a 5-day loading regimen in healthy, male and female volunteers. A total of 30 subjects, ages 18-45, will be enrolled in the study, allocated equally among 3 cohorts of 10 subjects each, 8 treated with active drug and 2 with placebo. Subjects in Cohorts 1 and 3 will receive an oral dose of 75 mg or 150 mg, respectively, of study medication daily for 14 days. Subjects in Cohort 2 will receive 150 mg daily for 5 days followed by 2 additional doses of 150 mg on Days 9 and 14. Subject participation will include a screening visit within 28 days of study entry, a 14 day in-patient treatment period, and a 14 day out-patient follow-up phase. Safety will be assessed by study personnel continually during the 14 day in-patient treatment period and the out-patient follow-up phase. Adverse events will be recorded for all subjects. Other safety measures include laboratory tests, electrocardiograms (ECGs), visual and neurological assessments, physical examinations, and vital signs. Study duration will be approximately 6 months. Subject participation duration will be 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 45 years of age (inclusive).
* Subject must be a healthy male or female volunteer (i.e., hematology, clinical chemistries and urinalysis tests must be within study-defined ranges. Clinical tests must be performed within 28 days of receiving first dose of study drug.
* Body Mass Index (BMI) must be between 18.0 and 30.0 kg/m^2 inclusive.
* Subject must be Tuberculin Skin Test/Purified Protein Derivative (TST/PPD) negative (within the previous 1 year) at Screening. The TST/PPD may be omitted if the subject presents written evidence of having a negative test during the previous 12 months.
* Subject must be able to give voluntary written informed consent before any study related procedure is performed.
* If female, has no childbearing potential or agrees to avoid becoming pregnant from the day of screening through their entire participation in the trial (Day 28) by using one of the following acceptable methods of birth control plus recommended use of a barrier method (condom) by the male partner (even if vasectomized):

  1. intrauterine contraceptive device
  2. diaphragm in combination with contraceptive jelly, cream, or foam
  3. spermicide
  4. abstinence
* Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy or status after hysterectomy.
* Hormonal contraceptives of any type or form (including oral, transdermal, vaginal or depot preparations) will not be allowed during the study.
* All female subjects of childbearing potential must have a negative serum pregnancy test at screening and within 24 hours of the first dose of study product.
* Male subjects must agree to use an acceptable barrier method for birth control (abstinence or use of a condom with spermicide) from screening through Study Day 28 and advise and recommend use of additional birth control to female sex partners throughout the study.
* Subject agrees not to donate blood during the study and up to 30 days after Study Day 28.
* Subject agrees to comply with all study requirements, including clinic house rules.

Exclusion Criteria:

* A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Principal Investigator (PI), would jeopardize the safety of the subject or impact the validity of the study results.
* Subject has been on an abnormal diet during the 4 weeks preceding the study. Abnormal diet is defined as a diet in which the subject has a significant change in eating habits (e.g., liquid diet only) and an unbalanced diet (e.g., protein only, high fat, low carbohydrate, etc.).
* Subject has received an investigational drug in a clinical trial within 30 days prior to study initiation.
* Subject has used any over-the-counter (OTC) medication, including vitamins and herbal supplements, within 7 days prior to Day 1 of the study, unless in the opinion of the PI, the substance would not likely impact on the conduct of this study, including pharmacokinetics (PK) of SQ109.
* Subject has used any prescription medication within 14 days prior to Day 1 of the study, or the use of hormonal preparations containing sex hormones within 30 days prior to Day 1 of the study.
* Subject has any current medical condition requiring treatment with medication, either prescription or OTC.
* Subject has been treated with any known CYP450 enzyme altering drugs such as azoles, antifungals, barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to Day 1 of the study.
* Subject has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody and/or a positive urine screen for alcohol or drugs of abuse.
* Subject has a baseline QTc interval >450 msec (males) or >470 msec (females) or a family history of prolonged QTc syndrome or premature cardiac death.
* Subject has Wolf Parkinson White Syndrome (WPW) or family history of WPW or a history of supra-ventricular tachycardias or syncope.
* Subject has lived with a person with active tuberculosis (TB) with the past 12 months or has traveled to an area of endemic TB within the past 12 months.
* Subject has an abnormal result on the Ishihara color test, the funduscopic exam, current optic neuritis or known retinal disease.
* Subject has an uncontrolled intercurrent illness (i.e., active infection) or fever (oral temperature greater than or equal to 100.0 degrees Fahrenheit or greater than or equal to 37.7 degrees Celsius).
* Subject has had major surgery within 4 weeks of study entry.
* Women who are pregnant or breastfeeding.
* Subject has donated blood within the past 30 days prior to Day 1 of the study.
* Subject has allergy to ethambutol or related compounds.
* Subject is an employee of or family member of an employee of Sequella, Quintiles, or DynPort Vaccine Company LLC (DVC).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability evaluated by a review of physical examinations, color and visual acuity tests, funduscopic examinations, neurological examinations, vital signs assessments, 12-lead ECGs, routine clinical laboratory tests, and AE assessments. | Duration of study.

SECONDARY OUTCOMES:
Serial blood samples for the measurement of the plasma levels of SQ109 will be collected. Pharmacokinetic variables will be assessed. | Days 1, 2, 3, 4, 5, 6, 7-13 (Cohorts 1 and 3), 9 and 10 (Cohort 2 only), 14, 15, 16, 17, 18, 21, and 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States